CLINICAL TRIAL: NCT06197776
Title: Investigation of Multi-omics Technique to Predict the Efficacy of Chemoradiotherapy Combined With Immunotherapy for Recurrent and/or Metastatic Nasopharyngeal Carcinoma
Brief Title: Investigation of Multi-omics Technique to Predict the Efficacy of Chemoradiotherapy Combined With Immunotherapy for r/m NPC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Professor, Sun Yat-sen University
Other Study IDs: multi-omics technique in NPC
Record Dates: First submitted 2023-11-26; First posted 2024-01-09 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Multi-omics Technique; Nasopharyngeal Carcinoma; Recurrent and Metastatic Nasopharyngeal Carcinoma; Efficacy of Chemoradiotherapy and Immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chemoradiotherapy combined with immunotherapy: Patients treated with chemoradiotherapy combined with immunotherapy
  Interventions: Drug: cisplatin-based chemoradiotherapy combined with immunotherapy

INTERVENTIONS:
Drug: cisplatin-based chemoradiotherapy combined with immunotherapy — Chemotherapy:cisplatin-based chemotherapy
  GP/TP/PF/TPF
  Choice of chemotherapy regimen is decided by patient's doctor in charge.
  Radiation: Intensity Modulated Radiation Therapy
  All target volumes will be outlined slice by slice on the axial contrast-enhanced CT with MR fusion images in the treatment planning system. The target volumes are defined in accordance with the International Commission on Radiation Units and Measurements Reports 83. The prescribed dose is 70-72 Gy to PTVp (Planning target volume of the primary tumor), 64-70 Gy to PTVn (Planning target volume of the lymph node),60- 64Gy to PTV1 (High-risk planning target volume), and 54-58 Gy to PTV2 (Low-risk planning target volume) in 30-32 fractions. The details of dose limits for organs at risk are based on the study 0225 from The Radiation Therapy Oncology Group (RTOG 0225).
  Immunotherapy:PD-1 blocking antibody

SUMMARY:
The observational clinical study will recruit 50 recurrent and/or metastatic nasopharyngeal carcinoma (r/mNPC) patients, to investigate the prediction values of multi-omics technique for the efficacy of chemoradiotherapy combined with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic nasopharyngeal carcinoma patients
* All genders，range from 18～70 years old
* ECOG score 0 ~ 1
* Inform consent form

Exclusion Criteria:

* Have or are suffering from other malignant tumors;
* Participating in other clinical trials;
* Drug or alcohol addition;
* Do not have full capacity for civil acts;
* Mental disorder;
* Pregnancy or lactation;
* Severe complication, eg, uncontrolled hypertension.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent or metastatic nasopharyngeal carcinoma patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3 years
  To investigate the multi-omics technique to predict the 3-year failure-free survival of chemoradiotherapy combined with immunotherapy for r/m NPC patients

SECONDARY OUTCOMES:
ctDNA | through study completion, an average of 6 months
  To show the changes of ctDNA during the treatment among these patients
Tumor mutation load at DNA level | through study completion, an average of 6 months
  To show the changes of tumor mutation load at DNA level during the treatment among these patients
RNA expression | through study completion, an average of 6 months
  To show the changes of RNA expression during the treatment among these patients

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn